CLINICAL TRIAL: NCT00513552
Title: Treatment of Crohn's Disease With an Antibiotic Regimen Directed Against Mycobacterium Avium Paratuberculosis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No patient
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Timothy Koch, Physician, Medstar Health Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-257; FDA IND 75,897
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Rifabutin; Clarithromycin; Clofazimine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antibiotics (Experimental): Antibiotics
  Interventions: Drug: Rifabutin, Clarithromycin, and Clofazimine

INTERVENTIONS:
Drug: Rifabutin, Clarithromycin, and Clofazimine — Rifabutin 150 mg by mouth twice daily, Clarithromycin 250 mg by mouth twice a day, and Clofazimine 100 mg by mouth each morning

SUMMARY:
Crohn's disease is a chronic inflammatory disorder of the gastrointestinal tract. The origin of Crohn's disease remains unknown and there is no curative therapy, either medical or surgical, for this gut disorder.

It is believed that an infectious agent is important in the development of Crohn's disease. The similarity of Crohn's disease to the animal form of ileitis, termed Johne's disease, supports the possibility that both disorders are caused by exposure to Mycobacterium avium paratuberculosis or MAP. Multiple investigators have demonstrated good clinical responses of patients with Crohn's disease to treatment with triple antibiotic therapy directed against mycobacterial infection.

The hypothesis of this protocol is that triple antibiotic therapy is useful as a medical therapy for patients with Crohn's disease. The aim of this study is to examine the response of patients with Crohn's disease who are not receiving therapy with biological agents to triple antibiotic therapy.

DETAILED DESCRIPTION:
Clinical remission will be determined by a decline in the Crohns disease activity index to <151; clinical improvement will be examined using the inflammatory bowel disease (IBD) quality of life questionnaire; and endoscopic improvement will be examined using a Crohn's disease endoscopic activity index. All individuals must have had colonoscopy within 3 months of enrollment. An estimated 20 individuals will be enrolled in this protocol. Each patient will be treated for 6 months with a combination of rifabutin, clarithromycin, and clofazimine. At the end of 6 months of treatment for each patient, the Crohns disease activity index will be recalculated, each patient will again complete the IBD quality of life questionnaire, and each patient will undergo repeat colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* This study will only include patients capable of providing informed consent, ages 18 and older.
* Patients must have a documented diagnosis of Crohn's disease and have had a colonoscopy with photographs within 3 months prior to randomization.
* All patients must have a CDAI of 220 or greater at enrollment.
* All females must be post-menopausal, surgically sterilized, or either abstain from sexual intercourse or use a non-hormonal method of birth control other than or in addition to oral contraceptive during the study and for 6 weeks after the end of the study.

Exclusion Criteria:

* Any patient with ulcerative colitis
* All women of child-bearing age must have a negative urine pregnancy test within 1 week prior to the initial clinic visit.
* Patients receiving a biological therapy for Crohn's disease including remicade
* Patients with a known allergy to any of the three antibiotics used in this protocol.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07 (Estimated); Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Clinical remission by a decline in Crohns disease activity index to <151 | 6 Months
  Percent <151
Clinical improvement using inflammatory bowel disease quality of life questionnaire | 6 Months
  Improvement in QOL life questionnaire
Endoscopic improvement using Crohn's disease endoscopic activity index | 6 Months
  Endoscopic appearance

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R Koch, MD, Principal Investigator — Medstar Health Research Institute

REFERENCES:
- [Background] Karp SM, Koch TR, Pang G. Is there a MAP (Mycobacterium Avium Subspecies Paratuberculosis) for treating Crohn's disease? Practical Gastroenterology 31(4):40-50, 2007.